CLINICAL TRIAL: NCT01044524
Title: An Open Label Study to Determine ADME of 14C Labeled SLV334 and Its Metabolites After Single Intravenous Dose Infusion
Brief Title: Study to Investigate ADME of 14C Labeled SLV334 After an i.v. Infusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S334.1.004; 2009-017406-37 (EudraCT Number); 01044524 (Other Grant/Funding Number: NCT/NIH)
Record Dates: First submitted 2009-12-11; First posted 2010-01-08 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Pharmacology, Clinical
Keywords: 14C labeled ADME (Aborption Distribution Metabolism and Elimination) study; Phase I

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SLV 334
  Interventions: Radiation: SLV 334

INTERVENTIONS:
Radiation: SLV 334 — 2000 mg via i.v. solution

SUMMARY:
This study will investigate the absorption, distribution, metabolism and excretion after giving 2000 mg 14C-SLV334 via a 1-hour infusion. The absolute bioavailability will also be determined.

ELIGIBILITY:
Inclusion Criteria healthy non-smoking subjects Exclusion Criteria QTc > 430 ms; positive drug screen

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Percentage excreted in urine and feces | 16 days
metabolic profile SLV334 | 16 days
AUC, CL, lambda z, Cmax, t1/2, tmax and Vss | 16 Days

SECONDARY OUTCOMES:
adverse events | 16 days
vital signs | 16 days
ECG | 16 days
Laboratory safety variables | 16 days
Physical examination | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Anita Vanderlaan, Study Director — Abbott Products
Locations (1):
- S334.1.004 - Site 1, Zuidlaren, Netherlands